CLINICAL TRIAL: NCT05905666
Title: Effectiveness of Health Education and Counseling on Stages of Change in Smoking Cessation Behavior, Smoking Decisional Balance, and Self-efficacy of Smoking Cessation: A Prospective Self-control Study
Brief Title: Health Education and Counseling in Smoking Cessation Behavior, Smoking Decisional Balance, and Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Chii Jeng, Professor, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGH-OP108004
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2019-08

CONDITIONS: Coronary Heart Disease; Smoking Cessation; Smoking Behaviors
Keywords: self-efficacy; counseling; health education; smoking cessation behavior
MeSH Terms: conditions — Coronary Disease; Smoking Cessation; Smoking; Health Education | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The research period was divided into a control stage (first to fourth week: standard of care) and the experimental stage (fifth to eighth week: health education and counseling). In the control stage, participants only received standard nursing care. In the experimental stage, intervention measures (health education and counseling) were implemented. The baseline data were the pretest data collected in the control stage. Four weeks later, a posttest was performed, namely the pretest of the experimental stage. Subsequently, 4 weeks of health education and counseling were introduced to smokers according to different stages. After 4 weeks of intervention, participants were asked to fill out the posttest questionnaire again to measure the stages of change for smoking cessation, smoking decisional balance, and self-efficacy of smoking cessation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self-controlled design (Experimental): The research period was divided into a control stage (first to fourth week: standard of care) and the experimental stage (fifth to eighth week: health education and counseling).
  Interventions: Behavioral: health education and counseling

INTERVENTIONS:
Behavioral: health education and counseling — In the control stage, participants only received standard nursing care. In the experimental stage, intervention measures (health education and counseling) were implemented. The baseline data were the pretest data collected in the control stage. Four weeks later, a posttest was performed, namely the pretest of the experimental stage. Subsequently, 4 weeks of health education and counseling were introduced to smokers according to different stages. After 4 weeks of intervention, participants were asked to fill out the posttest questionnaire again to measure the stages of change for smoking cessation, smoking decisional balance, and self-efficacy of smoking cessation.

SUMMARY:
Most male smokers with coronary heart disease resume smoking after hospital discharge. The main reason for failure to quit smoking is lack of motivation. However, few studies have used individual health education models to explore the effectiveness of smoking cessation according to the stage of change in smoking cessation behavior of patients. The purpose of this study was to examine the effectiveness of health education and counseling on the stages of change, smoking decisional balance, and self-efficacy of smoking cessation in smokers with no intention of quitting.

DETAILED DESCRIPTION:
Patients diagnosed with coronary heart disease by a medical center and smoked habitually were recruited as participants through convenience sampling. The research period was divided into a control stage (first to fourth week: standard of care) and the experimental stage (fifth to eighth week: health education and counseling). In the control stage, participants only received standard nursing care. In the experimental stage, intervention measures (health education and counseling) were implemented. The baseline data were the pretest data collected in the control stage. Four weeks later, a posttest was performed, namely the pretest of the experimental stage. Subsequently, 4 weeks of health education and counseling were introduced to smokers according to different stages. After 4 weeks of intervention, participants were asked to fill out the posttest questionnaire again to measure the stages of change for smoking cessation, smoking decisional balance, and self-efficacy of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with coronary heart disease by a medical center and smoked habitually

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of smoking decisional balance | The changes of smoking decisional balance was measured at the first week, 4th week and the 8th week.
  The Chinese version of the smoking decisional balance scale is used to measure the changes of smoking decisional balance.This scale encompassed six items, consisting of the pro and con dimensions.
Changes of self-efficacy of smoking cessation | The changes of self-efficacy of smoking cessation was measured at the first week, 4th week and the 8th week.
  The self-efficacy of smoking scale is used to measure the level of confidence to resist smoking. The scale comprised 14 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No